CLINICAL TRIAL: NCT00748943
Title: The Clinical Effects of a Mouthwash Containing Chlorine Dioxide on Oral Malodor and Salivary Periodontal and Malodorous Bacteria Using for 7days
Brief Title: Clinical and Microbiological Effects of a Mouthwash Containing Chlorine Dioxide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Kayoko Shinada/DDS, phD, Dept. of Oral health promotion, Tokyo medical and dental university
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2_Shinada; 2_Shinada
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Halitosis
Keywords: chlorine; dioxide; mouthwash; halitosis; bacteria; saliva
MeSH Terms: conditions — Halitosis | interventions — chlorine dioxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Chlorine Dioxide — Experimental mouthwash (ClO2 Fresh®) contained 0.16% sodium chlorite (NaClO2)
  Other Names: ClO2 Fresh®

SUMMARY:
Previous research has shown the oxidizing properties and microbiological efficacies of chlorine dioxide (ClO2). However, no clinical studies have investigated its microbiological efficacies on periodontal and malodorous bacteria. The aim of this study was to assess the inhibitory effects of a mouthwash containing ClO2 on morning oral malodor and on salivary periodontal and malodorous bacteria using for 7 days.

DETAILED DESCRIPTION:
Background: Previous research has shown the oxidizing properties and microbiological efficacies of chlorine dioxide (ClO2). Its clinical efficacies on oral malodor have been evaluated and reported, however, no clinical studies have investigated its microbiological efficacies on periodontal and malodorous bacteria. The aim of this study was to assess the inhibitory effects of a mouthwash containing ClO2 on morning oral malodor and on salivary periodontal and malodorous bacteria using for 7 days.

Methods: A randomized, double blind, crossover, placebo-controlled clinical trial was conducted among 15 healthy male volunteers, who were divided into 2 groups. In the first test phase, the group 1 subjects (N = 8) were instructed to rinse with the experimental mouthwash containing ClO2 twice per day for 7 days, and those in group 2 (N = 7) to rinse with the control (placebo) mouthwash without ClO2. In the second test, phase after a one week washout period, each group had used the opposite mouthwash for 7 days. At baseline and after 7 days, oral malodor was evaluated with OM, and concentrations of hydrogen sulfide (H2S), methyl mercaptan (CH3SH) and dimethyl sulfide ((CH3)2S), the main VSCs of human oral malodor, were evaluated with GC. Clinical outcome variables included plaque and gingival indices, and the Winkel Tongue Coating Index(WTCI). The samples of saliva were microbiologically investigated.

Outcome variables were compared by t-test and Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral malodor

Exclusion Criteria:

* Oral malodor caused by foods

Ages: 19 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Oral malodor | 7 days

SECONDARY OUTCOMES:
Periodontal bacteria | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kayoko Shinada, DDS,phD, Principal Investigator — Dept. of Oral health promotion, Tokyo medical and dental university

REFERENCES:
- [Derived] Shinada K, Ueno M, Konishi C, Takehara S, Yokoyama S, Zaitsu T, Ohnuki M, Wright FA, Kawaguchi Y. Effects of a mouthwash with chlorine dioxide on oral malodor and salivary bacteria: a randomized placebo-controlled 7-day trial. Trials. 2010 Feb 12;11:14. doi: 10.1186/1745-6215-11-14. PMID 20152022